CLINICAL TRIAL: NCT02786004
Title: Mammography Image Quality Assessment Reading NextGen Images for Screening and Diagnostic Use (MAGNIFI)
Brief Title: Image Quality Assessment for Screening and Diagnostic Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 124.03-2015-GES-0004
Record Dates: First submitted 2016-05-24; First posted 2016-05-30 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Breast Health
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Field Digital Mammography (Experimental): 2-dimensional breast imaging
  Interventions: Device: Full Field Digital Mammography
- Digital Breast Tomosynthesis (Experimental): 3-dimensional breast imaging
  Interventions: Device: Digital Breast Tomosynthesis

INTERVENTIONS:
Device: Full Field Digital Mammography
  Other Names: 2D Mammography
  Arms: Full Field Digital Mammography
Device: Digital Breast Tomosynthesis
  Other Names: DBT
  Arms: Digital Breast Tomosynthesis

SUMMARY:
This study is being conducted to determine the image quality of images using a new investigational medical imaging device.

ELIGIBILITY:
Inclusion Criteria:

1. Are women aged 40 years or older (≥40 years old);
2. Have had a FFDM (Full Field Digital Mammography) or DBT (Digital Breast Tomosynthesis) breast imaging exam within 30 days prior to enrollment;
3. Have breast sizes compatible with the dimensions of a 24x29 cm image detector without anatomical cut-off;
4. Are able to walk without assistive devices;
5. Are sterile; post-menopausal; or if of childbearing potential, have a negative pregnancy test or is willing to provide urine sample to confirm no pregnancy, within 30 days of imaging exam; and
6. Are willing to provide written informed consent to participate.

Exclusion Criteria:

1. Have been previously included in this study or are participating in another trial expected to interfere with study procedures or outcomes;
2. Have a history of breast biopsy, lumpectomy or mastectomy, or reconstruction on either breast;
3. Are currently lactating;
4. Are currently undergoing radiotherapy or chemotherapy , or have a history of prior radiotherapy treatment on either breast; or
5. If enrolled to the DBT (Digital Breast Tomosynthesis) cohort, have breast implants (breast implants are not exclusionary in the FFDM (Full Field Digital Mammography) cohort).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Schroeder, MD, Principal Investigator — Carolina Breast Imaging Specialists
Locations (1):
- Carolina Breast Imaging Specialist, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Field Digital Mammography: 2-dimensional breast imaging
  Full Field Digital Mammography
- Digital Breast Tomosynthesis: 3-dimensional breast imaging
  Digital Breast Tomosynthesis
Period: Overall Study
Arm/Group | Full Field Digital Mammography | Digital Breast Tomosynthesis
Started | 14 | 10
Completed | 14 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Field Digital Mammography | Digital Breast Tomosynthesis | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acceptable Overall Clinical Image Quality
Description: Overall clinical image quality was assessed by Mammography Quality Standards Act (MQSA) qualified radiologists ("readers"). Readers documented acceptability of FFDM and DBT image quality and image characteristics, as set for in the Guidance for Industry and FDA Staff - Class II Special Controls Guidance Document: Full Field Digital Mammography System (2012).
Time Frame: At enrollment completion approximately 3 months post initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Full Field Digital Mammography | Digital Breast Tomosynthesis
Number analyzed (Participants) | 14 | 9
Participants | 14 | 9

2. Secondary Outcome: Number of Subjects Experiencing a Device Related Adverse Events, Serious Adverse Event, Unanticipated Device Effect, and Device Defects by Overall Occurrence.
Description: Safety-related endpoint data (adverse events, serious adverse event, unanticipated device effect, and device defects) were monitored from all subjects for the duration of their participation. Results were summarized by cohort.
Time Frame: Through study completion, approximately 3 months
Population: Twenty-four subjects were enrolled into the study, of which 14 were enrolled into the FFDM cohort and 10 into the DBT cohort. One (1) subject was withdrawn from the DBT cohort but was followed for AE, SAE, and UADE for the duration of her participation.
Measure: Number; unit: participants
Groups:
- Full Field Digital Mammography: Subjects underwent two-dimensional breast imaging.
- Digital Breast Tomosynthesis: Subjects underwent three-dimensional breast imaging.
Arm/Group | Full Field Digital Mammography | Digital Breast Tomosynthesis
Number analyzed (Participants) | 14 | 10
participants
  Adverse Events | 0 | 0
  Serious Adverse Events | 0 | 0
  Unanticipated Device Effect | 0 | 0
  Device Defects | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the duration of subject participation in the study, which was approximately 2 months.
Arm/Group | Full Field Digital Mammography | Digital Breast Tomosynthesis
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 0/14 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No